CLINICAL TRIAL: NCT00501904
Title: Efficacy of Long- Versus Short-term Metformin Protocol in Infertile Anovulatory PCOS Patients
Brief Title: Metformin in Infertile PCOS Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/2006b
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Anovulation; Infertility; Metformin; PCOS; Treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Infertility | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Short protocol
  Interventions: Drug: Metformin
- Group B (Active Comparator): Long protocol
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Metformin, an oral biguanide administrated for treating type-2 diabetes mellitus, is a safe and effective drug recently experimented also in patients with polycystic ovary syndrome (PCOS). The administration of metformin induces ovulatory cycles in CC-resistant or -nonresistant patients with PCOS, and improves the ovulation rate as an additional treatment in women who received CC.

To date, it is unknown the best protocol for metformin administration. In particular, it is not known how long patients who ovulate under metformin should continue treatment before switching to second-line ovulation induction therapy. In this regard, in a recent study by the Kaplan-Meier survival analysis we demonstrated that the first pregnancy occurred late after metformin with an estimated median of seven months.

Based on these considerations, the aim of the present study will be to evaluate the clinical efficacy of metformin according to its duration of administration in infertile PCOS patients ovulating under treatment.

DETAILED DESCRIPTION:
Infertile PCOS patients having three ovulatory cycles under metformin, administered using tailored protocol, will be enrolled and randomized in two groups (groups A and B). Patients of group A will continue metformin administration for further three cycles followed by six months of progestogens cyclically administered, whereas patients of group B will continue metformin therapy for further nine cycles.

All patients eligible will undergo baseline assessment consisting of anthropometric, hormonal, and ultrasonographic evaluations. During the study, the clinical and reproductive outcomes, and the adverse experience will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant. Continuous variables will be analyzed with the unpaired t test and general linear model for repeated measures analysis with Bonferroni test for the post-hoc analysis as required. For categorical variables, the Pearson chi-square and Fisher's exact tests will be used. Cumulative pregnancy rate, our primary end-point, will be calculated by the Kaplan-Maier method, and the differences between the two groups will be assessed with the log-rank test. Cox proportional-hazards model will be used to calculate the hazard ratio for new pregnancy in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using NIH criteria)
* Anovulatory infertility (using WHO criteria)
* Ovulatory cycles under metformin (three cycles)

Exclusion Criteria:

* Age <18 or >35 years
* Severe obesity (BMI >35)
* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetic and anti-obesity drugs or other hormonal drugsPrevious use of ovulation induction agents
* Intention to start a diet or a specific program of physical activity
* Organic pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 12 months

SECONDARY OUTCOMES:
Ovulation rate Abortion rate Live-birth rate Adverse events | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Magna Graecia" of Catanzaro; Francesco Orio, MD, Principal Investigator — Department of Endocrinology, University "Federico II" of Naples; Achille Tolino, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Federico II" of Naples
Locations (1):
- Pugliese Hospital, Catanzaro, Catanzaro, CZ, Italy, Italy

REFERENCES:
- [Background] Palomba S, Orio F Jr, Falbo A, Russo T, Tolino A, Zullo F. Clomiphene citrate versus metformin as first-line approach for the treatment of anovulation in infertile patients with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Sep;92(9):3498-503. doi: 10.1210/jc.2007-1009. Epub 2007 Jun 26. PMID 17595241
- [Background] Palomba S, Orio F Jr, Falbo A, Manguso F, Russo T, Cascella T, Tolino A, Carmina E, Colao A, Zullo F. Prospective parallel randomized, double-blind, double-dummy controlled clinical trial comparing clomiphene citrate and metformin as the first-line treatment for ovulation induction in nonobese anovulatory women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Jul;90(7):4068-74. doi: 10.1210/jc.2005-0110. Epub 2005 Apr 19. PMID 15840746